CLINICAL TRIAL: NCT05675852
Title: Evaluation of Visual Parameters in Healthy and Visually Impaired Adults Using the Sweep and Oddball Technique Associated With Visual Evoked Potentials Captured by EEG
Brief Title: Evaluation of Visual Parameters by Visual Evoked Potentials Captured by EEG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: 2017%244
Record Dates: First submitted 2023-01-03; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Visual Neurosciences

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy participants: Healthy participants aged from 1 to 75 years old. All experiments conducted in this study will make use of the electroencephalogram (EEG) recording technique. Healthy participants cannot participate if they suffer from dermatosis on the scalp. There is no other contraindication to the practice of an EEG, which simply consists of recording the electrical activity of the brain on a trace, after application of a conductive gel on the scalp where sensors connected to a recording device are placed.
  We will collect the cerebral electrical response by the technique of steady state visual evoked potentials (SSVEP) which consists of presenting a visual stimulus periodically to interpret the EEG signal according to those variations.
  Interventions: Other: 68-electrode electroencephalography with steady state visual evoked potentials

INTERVENTIONS:
Other: 68-electrode electroencephalography with steady state visual evoked potentials — Electroencephalography is registered through a 68-electrode electroencephalography while stimuli will be presented at the centre of the screen at a distance of 150cm.
  The pattern of visual stimulation is based on the technique of steady state visual evoked potentials. These potentials consist of the presentation of a visual stimulus at a (relatively fast) periodic rate to produce an EEG signal over the occipital cortex exactly at the frequency of stimulation. By varying the value of a parameter of the stimulation (e.g. the contrast of the stimulus) varies. This variation makes it possible to determine the threshold value where an EEG response is perceived, and thus to evaluate visual parameters such as visual acuity, contrast sensitivity or recognition of more complex shapes.

SUMMARY:
This project will be based on an approach that has already proven itself in the field of the development of low-level visual functions such as visual acuity, vernier acuity and contrast sensitivity (Norcia & Tyler, 1985): scanning visual evoked potentials" (sVEP), a special case of steady-state visual evoked potentials (SSVEP). While SSVEPs consist of presenting a visual stimulus periodically, sVEPs are SSVEPs where the value of a parameter (e.g. the contrast of the stimulus) varies. This variation ("scanning") makes it possible to determine the threshold value where an electroencephalographic (EEG) response is perceived, and thus to evaluate visual parameters such as visual acuity, vernier acuity and contrast sensitivity. In this study we therefore record the amplitude of the EEG electrical signal during the presentation of low-level stimuli such as spatial frequency gratings or increasing or decreasing contrast.

ELIGIBILITY:
Inclusion Criteria:

* Absence of ocular pathologies except for refractive errors
* Absence of neurologic conditions

Exclusion Criteria:

* Participants using neurologic or psychiatric drugs
* Scalp pathology

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy participants to better understand visual neurosciences.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Threshold of visual recognition of low and high grade visual stimuli | 4 months
  Fast periodic visual stimulation using stimuli such as gratings, checkerboards, words and faces

CONTACTS AND LOCATIONS:
Locations (1):
- Institute Of NeuroSciences, Woluwe-Saint-Lambert, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No